CLINICAL TRIAL: NCT04143620
Title: Triple Procedure for Dense Cataractus Neovascular Glaucoma Patients
Acronym: NVG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shaaban Elwan, Assistant professor of ophthalmology, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minia University, NVG
Record Dates: First submitted 2019-10-27; First posted 2019-10-29 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-10

CONDITIONS: IOP Decreased; Visual Impairment
MeSH Terms: conditions — Ocular Hypotension; Vision Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Manegment of uncontrolled NVG patients with dense cataract
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neovascular glaucoma (Other): Neovascular glaucoma patients underwent triple procedure
  Interventions: Procedure: Procedure

INTERVENTIONS:
Procedure: Procedure — Triple procedure
  Other Names: Triple procedure

SUMMARY:
Background: One of the most difficult refractory glaucomas in treatment is the neovascular type and its association with dense cataract add to this difficulty. This study aimed to provide results of triple surgical treatment of such conditions.

Methods: A total of 12 eyes of 12 patients with dense cataractus NVG patients were included in this study. The patients mean age was 57.25 ± 5.9 years. The mean pre-operative intraocular pressure (IOP) was 47.25 ± 4.04 mmHg with maximum antiglaucoma therapy. The mean best corrected distant visual acuities (BCDVA) in log MAR was 2.13 ± 0.38. All the patients received intra-vitreal injection of 1.25 mg (0.05 ml) bevacizumab followed by phacoemulsification, pars plana vitrectomy (PPV) including pan-retinal photocoagulation (PRP), and assisted trabeculectomy with Mitomycin c (MMC). Mean IOP and BCDVA changes were the main outcome results of this study.

DETAILED DESCRIPTION:
Introduction Ocular ischemia due to diabetic retinopathy (DR) and central retinal vein occlusion (CRVO) are the most common causes that contribute to the development of neovascular glaucoma (NVG). Ischemic retina derived factors like vascular endothelial growth factor (VEGF) that can affect the anterior segment and initiates neovascularization in the iris (NVI), neovascularization in the angle (NVA). Aqueous outflow is obstructed when neovascular fibrous tissues block the trabecular meshwork and leads to synechial angle closure, thus NVG develops. Intraocular pressure (IOP) rise due to NVG lowers the ocular perfusion leading to further retinal ischemia, and this in turn induces more neovascularization. The management of NVG is very difficult thus; the conventional treatments such as antiglaucoma drugs, trabeculectomy, cyclophotocoagulation and cyclocryotherapy have poor success rates. It is very important to reduce the ischemic drive promptly for the treatment of NVG. Pan-retinal photocoagulation (PRP) is a mandatory and effective in resolving the ischemic condition and decreasing the vasoproliferative factors production.[ This management is particularly difficult in eyes with dense cataract. However, it is possible to overcome this difficulty by doing phacoemulsification and pars plana vitrectomy (PPV) + PRP. Moreover, phacoemulsification combined with PPV enables us to apply PRP from the posterior pole to the ora serrata peripherally. It has been known that Mitomycin C (MMC) increase the success rate of trabeculectomy in patients with NVG. Therefore, in the current study, we performed Intravitreal bevacizumab (IVB) injection, phacoemulsification, PPV + PRP and trabeculectomy augmented with subconjunctival injection of MMC.

The aim of this study is to evaluate safety and efficacy of this combined surgical procedure to alleviate retinal ischemia, reduce IOP, and improve visual acuity in dense cataractus NVG patients.

Subjects and Methods

Twelve eyes of 12 patients with NVG associated with dense cataract enough to obscure fundus visualization (7 males, 5 females) were included in the study in the period from July 2016 to August 2019 at Ophthalmology Department, Faculty of Medicine, Minia University. The patient's age ranged from 47 to 66 years with a mean age of 57.25 ± 5.9 years. The underlying cause for NVG was diabetes mellitus (DM) in 8 eyes (75%) and CRVO in 4 eyes (33.33%). Vitreous hemorrhage was present in half (50%) of the patients. The study was approved by the Local Ethical Review Committee and adhered to the tents of Declaration of Helsinki as well as all patients singed a written consent after discussion of the potential benefits and risks of this triple surgical procedures.

Preoperative examinations: Routine ophthalmological examinations were done after history taking including, age, sex, laterality, etiology of NVG and number of used anti-glaucoma drugs. The ocular examination includes estimation of visual acuity, IOP measurement with Goldman applanation tonometer, slit lamp examination of anterior segment, gonioscopy examination of angle of anterior chamber, biometry and ultrasonography. The demographic data were registered as in (Table 1).

Surgical procedures . In brief: - All procedures were done under peribulbar anesthesia with mild systemic sedation. IVB injection of 1.25 mg (0.05 ml) was given 2-6 days before surgery using a 27-gauge needle at the inferotemporal quadrant at 3.5-4.0 mm posterior to the limbus. Preoperative IV mannitol was given to all cases to lower IOP before surgery beside the full anti-glaucoma drugs including: topical Dorzolamide-Timolol combination, Brimonidine tartrate and oral Acetazolamide (250 mg) three times a day. Subconjunctival injection of MMC in a dose of 0.04mg/ml was done, and a period of 4 minutes was left before Conjunctival opening.

Fornix based Conjunctival incision was performed and a rectangular scleral flap of 3x4 mm was dissected. Separate temporal clear corneal incision phacoemulsification was done with intrabagal one-piece hydrophobic IOL implantation. Then, incision was closed with 10/0 nylon suture. This was followed by three ports 25-G PPV including core vitrectomy, injection of triamcinolone acetonide, induction of PVD, shaving of vitreous base, and dealing with any epiretinal membranes. PRP using diode endo-laser was done up to the far periphery (2000-3000 shots, duration 200 ms; power 400 mw). Fluid-air exchange was then performed and 20% SF6 was injected leaving 10 cc of gas to adjust pressure at the end of surgery. Then, the upper sclerotomies were sutured by vicryl 7/0 and the infusion cannula was left in place connected to the syringe of 20% SF6. Then, Healon was injected into the anterior chamber to maintain depth of anterior chamber and trabeculectomy by Kelly punch and peripheral iridectomy were done. Scleral flap was sutured by two 10/0 nylon sutures at the corners followed by watertight Conjunctival wound closure. More SF6 was injected to adjust IOP and the infusion cannula was removed, and its site was sutured with vicryl 7/0 suture. At the end of surgery, fluid was injected into the AC to test for filtration of bleb and to make sure that the conjunctiva was closed watertight. At last, triamcinolone acetonide subtenon injection was given to all eyes.

Post-operative management: The patients were prescribed prednisolone 1% (predfort, Alcon Co.) eye drops QID and tapered through 8 weeks, cyclopentolate 0.5 % TID, moxifloxacin 0.3 mg (Vigamox, Alcon Co.) eye drops QID for 2 weeks and ointment of tobramycin and dexamethasone at night for 4 weeks. Scheduled follow up visits were advised next postoperative day, one week, two weeks, monthly for three months, and then each three months for 2 years.

All patients underwent full ophthalmologic examination including BCDVA, IOP, gonioscopy, slit lamp examination, and dilated fundus examination. Antiglaucoma medications were prescribed if IOP was more than 21 mmHg. Baseline results and that of 1, 3 and 6 months, 1 and 2 years were included in the statistical analysis. This study main outcome measures were the mean BCDVA (log MAR), the mean IOP and the incidence of complications. Successful surgery was considered when the target IOP =21 mmHg was achieved without serious complications such as suprachoroidal hemorrhage, choroidal effusion, retinal detachment, endophthalmitis, phthisis bulbi, or persistent hypotony (IOP <5 mmHg). Complete success was considered when IOP of 6 -21 mmHg was achieved without any anti-glaucoma drugs, and qualified success when this target IOP was achieved with and without the use of anti-glaucoma drugs. Failure was defined as IOP >21 mmHg despite the use of maximum tolerated medications, hypotony, or the need for another glaucoma surgery.

Statistical analysis: Statistical analysis was performed with SPSS 19. Data were expressed as mean ± standard deviation (SD). Changes in the mean BCDVA and the mean IOP were compared for each follow up visit with baseline using paired t test and graphs construction done by using Graph Pad Prism 5 program. P value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients with uncontrolled angle closure dense cataractus NVG with maximum tolerated anti-glaucoma medications.

Exclusion Criteria:

* Excluded from this study eyes that had previous anti-glaucoma procedures, silicone oil filled eyes, previous buckle surgery or Conjunctival scaring from any cause, eyes with clear crystalline lens or faint cataract, eyes with corneal opacity, and eyes with visual acuity less than hand motion with good perception of light.

Ages: 47 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
BCDVA | 2 years
  Best corrected distant visual acuity
IOP | 2 years
  Intra-ocular pressure

SECONDARY OUTCOMES:
Post-operative complications | 2 years
  Post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Hossam M Moharram, MD, Study Chair — Minia University
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Results of the study
Supporting Information: CSR
Time Frame: 2 years
Access Criteria: study results

REFERENCES:
- [Derived] Moharram HM, Abd-Elhamid Mehany Elwan S, Nassar MM, Abdelkader MF. Triple Procedure for Dense Cataractous Neovascular Glaucoma Patients. J Ophthalmol. 2020 Jun 21;2020:1251203. doi: 10.1155/2020/1251203. eCollection 2020. PMID 32655940